CLINICAL TRIAL: NCT05890690
Title: Plasma Copeptin in Response to Oral Urea in Healthy Adults and Patients With Polyuria-polydipsia Syndrome: a Double-blind, Randomized, Placebo-controlled Cross-over Proof-of-concept and Pilot Study - The URANOS Study
Brief Title: Plasma Copeptin in Response to Oral Urea in Healthy Adults and Patients With Polyuria-polydipsia Syndrome
Acronym: URANOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2023-00751; kt23christcrain2
Record Dates: First submitted 2023-05-23; First posted 2023-06-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Arginine Vasopressin Deficiency; Primary Polydipsia
Keywords: diabetes insipidus; copeptin; oral urea
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Polydipsia, Psychogenic; Diabetes Insipidus | interventions — Blood Urea Nitrogen

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled cross-over proof-of-concept and pilot study
Who Masked: Participant, Investigator
Masking Description: Study staff and participants are blinded upon the nature of each study visit. The preparation of the study medication or placebo will be performed by unblinded study staff who is otherwise not involved in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Part 1 urea followed by placebo (Experimental): Participants will undergo a diagnostic test with a single weight-adapted dose of oral urea first. After a a wash-out phase of at least 3 days and not more than 28 days participants will undergo a second diagnostic test with a single weight-adapted dose of placebo.
  Interventions: Diagnostic Test: Urea; Diagnostic Test: Placebo
- Study Part 1 placebo followed by urea (Experimental): Participants will undergo a diagnostic test with a single weight-adapted dose of placebo first. After a a wash-out phase of at least 3 days and not more than 28 days participants will undergo a second diagnostic test with a single weight-adapted dose of urea.
  Interventions: Diagnostic Test: Urea; Diagnostic Test: Placebo
- Study part 2 Urea (Experimental): Participants will undergo a diagnostic test with a single weight-adapted dose of oral urea
  Interventions: Diagnostic Test: Urea

INTERVENTIONS:
Diagnostic Test: Urea — Diagnostic test with a single weight-adapted dose of oral urea dissolved in 200 ml water together with 5 g of lemon-lime flavor powder (containing maltodextrin and citric acid).
  The investigators will make use of the lemon-lime flavor to soften the bitter taste of urea.
  - Dose calculation: 0.5 g urea/kg body weight (rounded to no decimal places), with a minimal dose of 30g and a maximal dose of 45g.
Diagnostic Test: Placebo — Diagnostic test with a single weight-adapted dose of placebo dissolved in 200 ml water together with 5 g of lemon-lime flavor powder (containing maltodextrin and citric acid).
  The placebo will contain a mixture of bitter herbal substances to mimic the taste of urea.
  - Dose calculation: 22 ml of placebo containing 20 ml Ergytonyl®, 1 ml Carmol®, and 1 ml Bitter Liebe®.
  Arms: Study Part 1 placebo followed by urea; Study Part 1 urea followed by placebo

SUMMARY:
The aim of this study is to investigate whether oral urea stimulates copeptin release and, if so, whether it may provide a novel diagnostic test in the differentiation between AVP-D (Arginine vasopressin deficiency) and PP (primary polydipsia).

DETAILED DESCRIPTION:
This study consists of two parts, including healthy adults (study part 1 - proof of concept) and adults with an established diagnosis of PP or AVP-D (study part 2 - pilot study).

If the results of study part 1 suggest that oral urea is a potent stimulator of copeptin in healthy adults, study part 2 will be conducted, meaning that adults with an established diagnosis of PP or AVP-D will be included. If study part 1 demonstrates no relevant copeptin increase in response to oral urea, the study will be terminated thereafter and study part 2 will not be conducted.

ELIGIBILITY:
Healthy volunteers

Inclusion Criteria:

* Age ≥18 years
* Healthy with no medication except hormonal contraception

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Evidence of disordered drinking habits and diuresis defined as polyuria >50ml/kg body weight/24h and polydipsia >3l /24h
* Known allergy towards components of the study drink
* Pregnancy and breastfeeding
* Intention to become pregnant during the study
* Evidence of acute illness

Patients

Inclusion Criteria:

* Age ≥ 18 years
* Documented PP or AVP-D based on accepted diagnostic criteria, i.e., water deprivation test, hypertonic saline infusion test or arginine infusion test. Accordingly, patients must have evidence of disordered drinking habits and diuresis defined as polyuria >50ml/kg body weight/24h and polydipsia >3l /24h or must be on regular daily desmopressin medication

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Known allergy towards components of the study drink
* Pregnancy and breastfeeding
* Evidence of acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Difference in maximal increase in copeptin levels in plasma (pmol/l) | up to 6 time assessment until 150 minutes after baseline
  The difference in maximal increase in copeptin levels in plasma (pmol/l) within 150 minutes after oral intake of urea versus placebo, with the maximal increase being the difference between baseline copeptin values measured at the beginning of the test and maximal values measured between 30 and 150 minutes after ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland